CLINICAL TRIAL: NCT01266174
Title: Randomized, Double-blind, Parallel Trial Comparing the Effects of Eltoprazine (Adjunct to Anti-psychotics) With Placebo in Adults With Schizophrenia, in Improving One or More Dimensions of Cognitive Impairment Associated With Schizophrenia
Brief Title: Effects of Eltoprazine on Cognitive Impairment Associated With Schizophrenia (CIAS) in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amarantus BioScience Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGI12004
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Cognitive Impairment; Schizophrenia
Keywords: CIAS; Cognition; Schizophrenia; Eltoprazine
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia | interventions — eltoprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eltoprazine (Experimental): eltoprazine pill 2.5mg bid, eltoprazine pill 5mg bid, eltoprazine 7.5mg bid
  Interventions: Drug: Eltoprazine
- Placebo (Placebo Comparator): placebo pill 2.5mg bid, placebo pill 5mg bid, placebo 7.5mg bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltoprazine — Comparison of eltoprazine, dosed orally, for 8 weeks
  Other Names: eltropazine hydrochloride
  Arms: Eltoprazine
Drug: Placebo — Placebo to match eltoprazine
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if eltoprazine (as an adjunct to anti-psychotic medication) improves one or more aspects of cognitive impairment in adult schizophrenic patients.

DETAILED DESCRIPTION:
Schizophrenia is a common and highly disabling psychiatric disorder with population prevalence around 1%. The manifestations of schizophrenia fall into three major domains: 1) "positive" symptoms, such as delusions, hallucinations, and disorganization of behavior; 2) "negative symptoms," including social withdrawal, lack of motivation, and reduced expression of affect; and 3) cognitive dysfunction. Cognitive deficits are seen in most patients with schizophrenia.

Eltoprazine has agonist effects on both 5-HT1A and 5-HT1B receptors, which suggests that this drug may be useful for normalizing prefrontal cognitive abilities, reducing aggression and impulsivity, and improving cognitive function in schizophrenia.

This study will compare the effects of Eltoprazine (as an adjunctive treatment to anti-psychotics) with Placebo in Adults with a DSM IV/DSM IV TR diagnosis of schizophrenia, in potentially improving one or more dimensions of cognitive impairment associated with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Males and Females, 18-65 years of age, who meet the DSM-IV-TR for schizophrenia.

Must test negative for pregnancy at the time of enrollment based on a pregnancy test & agrees to use birth control during study.

Performance less than the max cutoff (in parentheses) for ONE of the following MCCB tests: i) Letter-number span (20); ii) HVLT total (31); and iii) CPT d-prime (3.47) BPRS Hallucinatory Behavior or Unusual Thought Content item scores ≤ 5

BPRS Conceptual Disorganization item score ≤ 4

Simpson-Angus Scale total score ≤ 6

CDRS total score ≤ 10

Able to complete the baseline MCCB validly as assessed by tester

WTAR raw score ≥ 6

Be treated with one of the following second generation antipsychotics: risperidone, olanzapine, quetiapine, asenapine, iloperidone or paliperidone for the previous two months, with no change in dose in the last month, or with injectable depot antipsychotics (fluphenazine, haloperidol decanoate, risperdal Consta or paliperidone sustenna) with no change in last 3 months

Laboratory results must show no clinically significant abnormalities.

Must have an ECG with QTc measurement performed at Screening that is not clinically significant.

Must have a negative drug screen.

Exclusion Criteria:

Current treatment with one of the following antipsychotics: clozapine, aripiprazole, lurasidone or ziprasidone.

Current treatment with any anti-cholinergic drug in doses above 2 mg daily for benztropine, 5 mg per day for trihexyphenidyl, and 50 mg day for diphenhydramine.

Current treatment with benzodiazepines in doses above 10 mg of diazepam (or the equivalent of another drug).

Patients with a DSM-IV diagnosis of alcohol or substance abuse within the last month or a DSM-IV diagnosis of alcohol or substance dependence within the last 6 months.

Have a significant suicide attempt within one year of Visit 1, answered yes to question 3, 4 or 5 on the C-SSRS at Visit 1,or are currently at risk of suicide in the opinion of the Investigator.

Patients with a hx of significant head injury/trauma. Patients with a clinically significant neurological, metabolic,hepatic, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorder. Insulin-dependent diabetics who are clinically stable and whose baseline fasting glucose is 200 or less may be included.

Clinically significant abnormalities in PE, ECG, or lab assessments. Clinically significant renal disease (e.g. chronic renal insufficiency with GFR <60, inflammatory disease requiring medication, acute renal failure).

Pregnant women or women of child-bearing potential, who are either not surgically-sterile or using appropriate methods of birth control.

Women who are breast-feeding Have a TSH level consistent with hyperthyroidism or hypothyroidism. Patients previously diagnosed with hyperthyroidism or hypothyroidism, who have been treated on a stable dose of thyroid supplement for at least the past 3 months, and who are clinically and chemically euthyroid will be allowed to participate in the study.

Have significant prior or current medical conditions that, in the judgment of the investigator, could be exacerbated by or compromised by study drug.

Have any medical condition that would increase sympathetic nervous system activity markedly.Patients who are taking a medication on a daily basis (for example, albuterol, inhalation aerosols, pseudoephedrine), that has sympathomimetic activity can be enrolled.

Used MAOIs during the 2 weeks (14 days) prior to Baseline. Have used any SSRI, a 5HT1A agonist or other serotonin-mediated treatment for any reason during the 4 weeks prior to Baseline.

Have current hypertension despite treatment. Have received treatment within the last 60 days with a drug that has not received regulatory approval for any indication at the time of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery (MCCB) | At Baseline and every 4 weeks
  Assessment of cognitive effects over time measured suing the MCCB battery

SECONDARY OUTCOMES:
Continuous Performance Test-AX Version (CPT-AX) | At Baseline and every 4 weeks
  Assessment of Cognitive effects over time measured using the Continuous Performance Test (AX version)
N-Back | At Baseline and every 4 weeks
  Assessment of Cognitive effects over time measured using the N-Back Working Memory Test
Brief Psychiatric Rating Scale (BPRS) | At Baseline and every 2 weeks
Calgary Depression Scale (CDS) | At Baseline and every 2 weeks
Scale for Assessment of Negative Symptoms (SANS) | At Baseline and every 2 weeks
Simpson-Angus Extrapyramidal Symptom Rating Scale (SAS) | At Baseline and every 2 weeks
Abnormal Involuntary Movement Scale (AIMS) | At Baseline and every 2 weeks
Barnes Akathisia Scale (BAS) | At Baseline and every 2 weeks
Columbia Suicide Severity Rating Scale (C-SSRS) | At baseline and end of study; every two weeks if there is a change in the CDRS suicidality rating to a score of 2 or 3

CONTACTS AND LOCATIONS:
Overall Officials: John G Csernansky, MD, Principal Investigator — NortWestern University Feinberg School of Medicine
Locations (6):
- United States (6):
  - Veteran's Administration of Greater Los Angeles, Los Angeles, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Maryland Psychiatric Research Center, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Research Foundation for Mental Hygiene, Inc., New York, New York
  - Duke University School of Medicine, Durham, North Carolina